CLINICAL TRIAL: NCT04431986
Title: Association Between Emergency Room Evaluation and Recommendations Tool (ER2) Frailty Levels and Incident Adverse Health Events in Older Community Dwellers: Results of the NuAge Study
Brief Title: ER2 Frailty Levels and Incident Adverse Health Events in Older Community Dwellers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Cyrille Launay, Principal Investigator, Jewish General Hospital
Other Study IDs: 2021-2432
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Frailty; Emergencies; Aging
MeSH Terms: conditions — Frailty; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NuAge participants: All Individuals of the NuAge study who agreed to be part of the NuAge Database for future research purposes
  Interventions: Other: No intervention: secondary use of a database

INTERVENTIONS:
Other: No intervention: secondary use of a database — Statistical analyses

SUMMARY:
Older adults' health and functional status are heterogeneous because of the various cumulative effects of chronic diseases and physiologic decline, contributing to a vicious cycle of increased frailty 1-4. Thanks to advances in medicine and hygiene, a growing number of older adults spend more years with a greater range of chronic diseases causing disability but not mortality 5. Health systems need to face this new challenge 4,5. Quantification of frailty and its association with the occurrence of incident adverse health events (i.e., functional decline, unplanned hospitalizations) is crucial to understand how health systems may efficiently respond to this situation 6. This study aims to examine the association of the ER2 tool score and its stratification in three levels for incident adverse health events in older community dwellers and to compare this association with three validity frailty indexes which are the Cardiovascular Health Study (CHS) frailty index, Study of Osteoporotic Fracture (SOF) index and Rockwood frailty index.

ELIGIBILITY:
Inclusion Criteria:

* All enrolled participants of NuAge Study who agreed to be part of the NuAge Database and Biobank for future research purposes

Exclusion Criteria:

* Missing data
* Participants' refusal to use their data for a purpose not identified during their recruitment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals eligible for this study will be participants of the NuAge study who agreed to be part of the NuAge Database and Biobank for future research purposes
Sampling Method: Non-Probability Sample
Enrollment: 1741 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
ER2 | 4 years
  6-item questionnaire determining a stratification of frailty risk in three levels (Low, moderate, high)
SOF index | 4 years
  index with 3 items determining a level of frailty from 0 (patient is vigorous) to 1 (patient is pre-frail)
CHS index | 4 years
  index with 5 items determining a level of frailty from 0 component positive (patient is vigorous), 1 or 2 positive components (patient is in an intermediate stage) to 3 or more positive components (patients is frail)
Rockwood index | 4 years
  index determining a level of frailty from 0 to 17 (less than 5: patient is vigorous, between 6 and 11 patient is apparently vulnerable and above 12 patient is in severe frailty)
Physical functional decline | 4 years
  annual variation of physical functional score available in the Nuage database
Falls | 4 years
  presence or absence of falls, information available in the Nuage database
Hospitalizations | 4 years
  presence or absence of hospitalizations, information available in the Nuage database
Mortality | 4 years
  death of the participant, information available in the Nuage database

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille Launay, MD, Principal Investigator — Jewish General Hospital

IPD SHARING:
Plan to Share IPD: No
The databank property is not ours. We do not have the right to share IPD.